CLINICAL TRIAL: NCT01602224
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Phase 2 Study of Tabalumab in Combination With Bortezomib and Dexamethasone in Patients With Previously Treated Multiple Myeloma
Brief Title: A Study of Tabalumab (LY2127399) in Participants With Previously Treated Multiple Myeloma (MM)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 14199; H9S-MC-JDCG (Other: Eli Lilly and Company)
Record Dates: First submitted 2012-05-16; First posted 2012-05-18 (Estimated); Results first posted 2018-08-15 (Actual); Last update posted 2019-10-08 (Actual); Status verified 2019-09

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Dexamethasone; Bortezomib; tabalumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 100 mg Tabalumab+Dexamethasone (Dex)+Bortezomib (BTZ) (Experimental): Tabalumab 100 milligram (mg) administered once intravenously (IV) over 30 minutes on Day 1 every 21 days for 8 cycles.
  Dexamethasone 20 mg administered once orally on Days 1, 2, 4, 5, 8, 9, 11 and 12 every 21 days for 8 cycles.
  Bortezomib 1.3 milligram per square meter (mg/m^2) administered once subcutaneously (SQ) on Days 1, 4, 8 and 11 every 21 days for a minimum 8 cycles.
  All treatment may continue past 8 cycles.
  Interventions: Drug: Dexamethasone; Drug: Bortezomib; Biological: Tabalumab
- 300 mg Tabalumab+Dexamethasone+Bortezomib (Experimental): Tabalumab 300 mg administered once IV over 30 minutes on Day 1 every 21 days for 8 cycles.
  Dexamethasone 20 mg administered orally on Days 1, 2, 4, 5, 8, 9, 11 and 12 every 21 days for a minimum 8 cycles.
  Bortezomib 1.3 mg/m^2 administered once SQ on Days 1, 4, 8 and 11 every 21 days for 8 cycles.
  All treatment may continue past 8 cycles.
  Interventions: Drug: Dexamethasone; Drug: Bortezomib; Biological: Tabalumab
- Placebo Comparator: Placebo + Dexamethasone + Bortezomib (Placebo Comparator): Placebo administered once IV on Day 1 every 21 days for 8 cycles.
  Dexamethasone 20 mg administered once orally on Days 1, 2, 4, 5, 8, 9, 11 and 12 every 21 days for a minimum 8 cycles.
  Bortezomib 1.3 mg/m^2 administered once SQ on Days 1, 4, 8 and 11 every 21 days for 8 cycles.
  All treatment may continue past 8 cycles.
  Interventions: Drug: Placebo; Drug: Dexamethasone; Drug: Bortezomib

INTERVENTIONS:
Drug: Placebo — Administered IV
  Arms: Placebo Comparator: Placebo + Dexamethasone + Bortezomib
Drug: Dexamethasone — Administered orally
Drug: Bortezomib — Administered SQ
Biological: Tabalumab — Administered IV
  Other Names: LY2127399
  Arms: 100 mg Tabalumab+Dexamethasone (Dex)+Bortezomib (BTZ); 300 mg Tabalumab+Dexamethasone+Bortezomib

SUMMARY:
The purpose of this study is to evaluate an investigational drug called tabalumab in participants with Multiple Myeloma (MM) who have tried at least one other therapy in the past. Tabalumab will be given in combination with standard doses of two other drugs that are often used to treat MM. Study doctors will collect information about the effectiveness and side effects of this therapy.

ELIGIBILITY:
Inclusion Criteria:

* Have symptomatic and/or progressive MM that was previously treated with at least 1 and no more than 3 prior lines of therapy
* Have measurable disease
* Have given written informed consent prior to any study-specific procedures
* Have adequate organ function
* Treatment with prior autologous transplant is permitted

Exclusion Criteria:

* Are enrolled in or discontinued from a clinical trial of any drug or device within 21 days prior to the first dose of assigned study treatment
* Have had less than a minimal response or have had progressive disease within 60 days of most recent therapy with a proteasome inhibitor
* Plan to proceed to autologous transplant for consolidation after participation in this trial
* Have an active infection or ongoing treatment for systemic infection ("ongoing treatment" does not include prophylactic anti-infectives),, chest x-ray suggestive of tuberculosis, or history/risk of chronic/latent infection that may reactivate in the presence of study therapy
* Have any of the following:

  * positive test results for human immunodeficiency virus (HIV)
  * positive test for hepatitis B, defined as positive for hepatitis B surface antigen (HBsAg+), OR positive for anti-hepatitis B core antibody AND positive for hepatitis B deoxyribonucleic acid (HBV DNA), OR positive for anti-hepatitis B surface antibody (HBsAb+) AND positive for hepatitis B deoxyribonucleic acid (HBV DNA)
  * positive test results for hepatitis C virus (HCV), defined as positive for hepatitis C antibody (HepCAb) AND confirmed positive via the hepatitis C recombinant immunoblot assay
* Have had significant allergy to human/humanized monoclonal antibodies that, in the opinion of the investigator, poses an unacceptable risk to the participants
* Have known hypersensitivity or contraindication to any of the study therapies or excipients
* Prior allogeneic hematopoietic stem cell transplant
* Prior therapy with experimental agents targeting B-cell activating factor (BAFF), including LY2127399
* Have corrected QT (QTc) interval >500 millisecond (msec) on baseline 12-lead electrocardiogram (ECG)
* Have Waldenstrom's macroglobulinemia
* History of malignancy with adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, in situ breast cancer, in situ prostate cancer, are eligible regardless of the time of diagnosis/treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2012-07; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (57):
- United States (14):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tucson, Arizona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fullerton, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Los Angeles, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Santa Barbara, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Grand Junction, Colorado
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Atlanta, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Indianapolis, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cedar Rapids, Iowa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Iowa City, Iowa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ashland, Kentucky
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Boston, Massachusetts
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Omaha, Nebraska
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Albuquerque, New Mexico
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Salt Lake City, Utah
- Brazil (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Campinas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Porto Alegre
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., São Paulo
- Canada (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Calgary, Alberta
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vancouver, British Columbia
- France (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lille
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nantes
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nîmes
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Paris
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tours
- Germany (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bamberg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cologne
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Heidelberg
- Greece (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ampelokipoi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Athens
- Italy (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bari
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Catania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Florence
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Milan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rome
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Torino
- Mexico (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mexico City
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Toluca
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rotterdam, Netherlands
- Poland (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Krakow
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lublin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Warsaw
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wroclaw
- South Korea (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Goyang-si
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seoul
- Spain (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Badalona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Barcelona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Madrid
- Taiwan (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Neihu Taipei
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Taipei
- Turkey (Türkiye) (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Izmir
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Melikgazi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sihhiye
- United Kingdom (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Headington, Oxford
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sutton, Surrey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Birmingham
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., London
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Manchester

IPD SHARING:
Plan to Share IPD: Yes
Lilly provides access to the individual patient data from studies on approved medicines and indications as defined by the sponsor specific information on ClinicalStudyDataRequest.com.
  This access is provided in a timely fashion after the primary publication is accepted. Researchers need to have an approved research proposal submitted through ClinicalStudyDataRequest.com. Access to the data will be provided in a secure data sharing environment after signing a data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Completers are defined as participants who died or had disease progression or completed treatment or did not complete treatment and were followed for survival data.
Groups:
- 100 mg Tabalumab+Dexamethasone+Bortezomib: Tabalumab 100 milligram (mg) administered once intravenously (IV) over 30 minutes on Day 1 every 21 days for 8 cycles.
  Dexamethasone 20 mg administered once orally on Days 1, 2, 4, 5, 8, 9, 11 and 12 every 21 days for 8 cycles.
  Bortezomib (BTZ) 1.3 milligram per square meter (mg/m^2) administered once subcutaneously (SQ) on Days 1, 4, 8 and 11 every 21 days for 8 cycles.
- 300 mg Tabalumab+Dexamethasone+Bortezomib: Tabalumab 300 mg administered once IV over 30 minutes on Day 1 every 21 days for 8 cycles.
  Dexamethasone 20 mg administered orally on Days 1, 2, 4, 5, 8, 9, 11 and 12 every 21 days for 8 cycles.
  Bortezomib 1.3 mg/m^2 administered once SQ on Days 1, 4, 8 and 11 every 21 days for 8 cycles.
- Placebo Comparator: Placebo + Dexamethasone + Bortezomib: Placebo administered once IV on Day 1 every 21 days for 8 cycles.
  Dexamethasone 20 mg administered once orally on Days 1, 2, 4, 5, 8, 9, 11 and 12 every 21 days for 8 cycles.
  Bortezomib 1.3 mg/m^2 administered once SQ on Days 1, 4, 8 and 11 every 21 days for 8 cycles.
Period: Overall Study
Arm/Group | 100 mg Tabalumab+Dexamethasone+Bortezomib | 300 mg Tabalumab+Dexamethasone+Bortezomib | Placebo Comparator: Placebo + Dexamethasone + Bortezomib
Started | 74 | 74 | 72
Received at Least 1 Dose of Study Drug | 73 | 74 | 72
Completed | 66 | 66 | 66
Not Completed | 8 | 8 | 6
Not completed — Adverse Event | 0 | 1 | 0
Not completed — Investigator Decison | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — Protocol Violation | 0 | 1 | 0
Not completed — Sponsor Decision | 2 | 3 | 2
Not completed — Withdrawal by Subject | 5 | 3 | 3

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- 100 mg Tabalumab+Dexamethasone+Bortezomib: Tabalumab 100 milligram (mg) administered once intravenously (IV) over 30 minutes on Day 1 every 21 days for 8 cycles.
  Dexamethasone 20 mg administered once orally on Days 1, 2, 4, 5, 8, 9, 11 and 12 every 21 days for 8 cycles.
  Bortezomib 1.3 milligram per square meter (mg/m^2) administered once subcutaneously (SQ) on Days 1, 4, 8 and 11 every 21 days for 8 cycles.
- Total: Total of all reporting groups
Arm/Group | 100 mg Tabalumab+Dexamethasone+Bortezomib | 300 mg Tabalumab+Dexamethasone+Bortezomib | Placebo Comparator: Placebo + Dexamethasone + Bortezomib | Total
Number analyzed (Participants) | 74 | 74 | 72 | 220
Age, Continuous [Median (Standard Deviation); unit: years] | 63.2 (11.01) | 65.7 (9.11) | 65.4 (9.50) | 64.8 (9.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 37 | 32 | 113
  Male | 30 | 37 | 40 | 107
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 3 | 5 | 12
  Not Hispanic or Latino | 39 | 50 | 35 | 124
  Unknown or Not Reported | 31 | 21 | 32 | 84
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 1 | 2 | 6
  Asian | 14 | 18 | 13 | 45
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 2 | 2 | 5
  White | 56 | 53 | 53 | 162
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 2 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 11 | 9 | 9 | 29
  United Kingdom | 5 | 7 | 4 | 16
  Spain | 8 | 5 | 8 | 21
  Greece | 6 | 7 | 9 | 22
  Canada | 2 | 2 | 0 | 4
  South Korea | 6 | 9 | 8 | 23
  Netherlands | 0 | 0 | 1 | 1
  Turkey | 6 | 7 | 4 | 17
  Taiwan | 7 | 6 | 5 | 18
  Brazil | 4 | 2 | 5 | 11
  Poland | 4 | 13 | 7 | 24
  Italy | 7 | 2 | 3 | 12
  Mexico | 3 | 1 | 2 | 6
  France | 3 | 3 | 6 | 12
  Germany | 2 | 1 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: PFS is defined as the time from date of first dose to the first observation of disease progression or death due to any cause. If a participant does not have a complete baseline disease assessment, then the PFS time is censored at the enrollment date, regardless of whether or not objectively determined disease progression (Increase of > 25% from lowest response in serum M component, urine M component, bone marrow plasma cell percentage, development of bone lesions) or death has been observed for the participant. If a participant is not known to have died or have objective progression as of the data inclusion cutoff date for the analysis, the PFS time is censored at the last complete objective progression-free disease assessment date.
Time Frame: Baseline up to Objective Disease Progression or Death From Any Cause (assessed up to 9 months)
Population: All randomized participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | 100 mg Tabalumab+Dexamethasone+Bortezomib | 300 mg Tabalumab+Dexamethasone+Bortezomib | Placebo Comparator: Placebo + Dexamethasone + Bortezomib
Number analyzed (Participants) | 74 | 74 | 72
months | 6.6 [5.6 to 8.5] | 7.5 [5.8 to 9.3] | 7.6 [6.5 to 9.3]

2. Secondary Outcome: Overall Survival
Description: Overall survival is the duration from enrollment to death from any cause. For participants who were alive, overall survival was censored at the last contact.
Time Frame: Baseline to Death From Any Cause (assessed up to 19 months)
Population: All randomized participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | 100 mg Tabalumab+Dexamethasone+Bortezomib | 300 mg Tabalumab+Dexamethasone+Bortezomib | Placebo Comparator: Placebo + Dexamethasone + Bortezomib
Number analyzed (Participants) | 74 | 74 | 72
months | NA [19.1 to NA] — Medians were not reached for timeframe | NA [NA to NA] — Medians were not reached for timeframe | NA [18.6 to NA] — Medians were not reached for timeframe

3. Secondary Outcome: Time to First Skeletal-Related Event (SRE)
Description: Time to first SRE is defined as time from randomization to any one of the following related to multiple myeloma: New Pathological Fracture, Spinal Cord Compression, Surgery to the Bone, Radiation to the Bone collected until participant death, study closure or lost to follow up. Participants not known to have had an SRE at the time of the analysis were censored at the date of their last complete documented assessment for SRE.
Time Frame: Baseline to Date of First Skeletal Related Event (assessed up to 19 months)
Population: All randomized participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | 100 mg Tabalumab+Dexamethasone+Bortezomib | 300 mg Tabalumab+Dexamethasone+Bortezomib | Placebo Comparator: Placebo + Dexamethasone + Bortezomib
Number analyzed (Participants) | 74 | 74 | 72
months | NA [NA to NA] — Medians were not reached for timeframe | NA [19.8 to NA] — Medians were not reached for timeframe | NA [NA to NA] — Medians were not reached for timeframe

4. Secondary Outcome: Number of Participants With >30% Reduction in Brief Pain Inventory (BPI) - Worst Pain Score
Description: BPI is assessed by 7 questions rated "0" for "no pain" and higher numbers indicated more pain.
Time Frame: Baseline through End of Treatment (19 months)
Population: All randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | 100 mg Tabalumab+Dexamethasone+Bortezomib | 300 mg Tabalumab+Dexamethasone+Bortezomib | Placebo Comparator: Placebo + Dexamethasone + Bortezomib
Number analyzed (Participants) | 74 | 74 | 72
Participants | 37 | 30 | 30

5. Secondary Outcome: Time to Progression (TTP)
Description: Time to progression is defined as the time from the date of randomization to the date of first observed objective progression or death due to study disease. Time to progression will be censored as for PFS for those participants not known to have progressed or that died from other causes.
Time Frame: Baseline to Objective Disease Progression or Death (assessed up to 9 months)
Population: All randomized participants, with 79 participants censored.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | 100 mg Tabalumab+Dexamethasone+Bortezomib | 300 mg Tabalumab+Dexamethasone+Bortezomib | Placebo Comparator: Placebo + Dexamethasone + Bortezomib
Number analyzed (Participants) | 74 | 74 | 72
months | 6.6 [5.9 to 9.3] | 8.2 [6.4 to 11.2] | 8.1 [6.9 to 9.5]

6. Secondary Outcome: Duration of Response (DoR)
Description: DOR is measured by the International Myeloma Working Group Uniform Response Criteria: from the date of first evidence of a confirmed response to the date of objective progression or the date of death due to any cause, whichever is earlier. If a responder is not known to have died or have objective progression as of the data inclusion cutoff date, the DOR time will be censored at the last complete objective progression-free disease assessment date. Progressive disease is an increase of 25% from baseline in Serum M, Urine M, bone marrow plasma cell increase of 10 %, development of new bone lesions, development of new soft tissue plasmacytomas or bone lesions, hypercalcemia >11.5 milligrams per deciliter, decrease in hemoglobin of 2 grams per deciliter, rise in serum creatinine by 2 mg/deciliter.
Time Frame: Time from Response to Objective Disease Progression (assessed up to 38 months)
Population: All randomized participants who received at least 1 dose of study drug and had a response.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | 100 mg Tabalumab+Dexamethasone+Bortezomib | 300 mg Tabalumab+Dexamethasone+Bortezomib | Placebo Comparator: Placebo + Dexamethasone + Bortezomib
Number analyzed (Participants) | 43 | 44 | 44
months | 7.9 [6.0 to 11.6] | 8.6 [6.5 to 10.7] | 7.7 [5.8 to 13.1]

7. Secondary Outcome: Time to Next Treatment (TNT)
Description: TNT is defined as the time from the date of randomization to the date of initiation of the first poststudy treatment course of anticancer therapy or death from any cause. Time to next treatment will be censored at the date of the last visit for participant who did not initiate additional anticancer therapy.
Time Frame: Baseline to Initiation of New Cancer Treatment or Death From Any Cause (18 Months)
Population: All randomized participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | 100 mg Tabalumab+Dexamethasone+Bortezomib | 300 mg Tabalumab+Dexamethasone+Bortezomib | Placebo Comparator: Placebo + Dexamethasone + Bortezomib
Number analyzed (Participants) | 74 | 74 | 72
months | 10.1 [7.0 to 11.9] | 9.9 [6.8 to 14.8] | 11.7 [7.8 to 17.5]

8. Secondary Outcome: Pharmacokinetics (PK): Maximum Concentration (Cmax) of Tabalumab
Description: Maximum Concentration (Cmax) of Tabalumab.
Time Frame: Cycle (C)1 Day (D)1: Predose, 3O minutes, 2 hours Postdose; C1 D4, 8, 11: Predose, (D11 only, 30 minutes Postdose); C2 and C6-C10 D1: Predose and immediately Postdose; C2 D 4, 8, 11: Anytime
Population: All randomized participants who received at least 1 dose of study drug and evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms per milliliter
Arm/Group | 100 mg Tabalumab+Dexamethasone+Bortezomib | 300 mg Tabalumab+Dexamethasone+Bortezomib
Number analyzed (Participants) | 68 | 71
micrograms per milliliter
  Cycle 1 | 38.0 (39) | 103 (43)
  Cycle 2: number analyzed (Participants) | 63 | 68
  Cycle 2 | 47.9 (51) | 131 (40)
  Steady State (Cycle 6-10) | 69.0 (51) | 189 (54)

9. Secondary Outcome: PK: Time to Maximum Plasma Concentration (Tmax) of Tabalumab
Time Frame: C1 D1: Predose, 3O minutes, 2 hours Postdose; C1 D4, 8, 11: Predose, (D11 only, 30 minutes Postdose); C2 and C6-C10 D1: Predose and immediately Postdose; C2 D 4, 8, 11: Anytime
Population: All randomized participants who received at least 1 dose of study drug with evaluable PK values.
Measure: Mean (95% Confidence Interval); unit: hours
Arm/Group | 100 mg Tabalumab+Dexamethasone+Bortezomib | 300 mg Tabalumab+Dexamethasone+Bortezomib
Number analyzed (Participants) | 73 | 74
hours
  Cycle 1 | 1.5 [0.75 to 503.75] | 1.58 [0.92 to 162.58]
  Cycle 2 | 0.92 [0.47 to 503.77] | 0.76 [0.5 to 503.58]
  Steady State (Cycle 6-10): number analyzed (Participants) | 47 | 74
  Steady State (Cycle 6-10) | 0.75 [0.338 to 9.92] | 0.73 [0 to 1.75]

10. Secondary Outcome: PK: Area Under the Curve Over the Dosing Interval (AUC-T) for Tabalumab
Time Frame: as for outcome 9
Population: All randomized participants who received at least 1 dose of study drug and had evaluable PK parameters.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms times hour per milliliter
Arm/Group | 100 mg Tabalumab+Dexamethasone+Bortezomib | 300 mg Tabalumab+Dexamethasone+Bortezomib
Number analyzed (Participants) | 68 | 71
micrograms times hour per milliliter
  Cycle 1 | 7790 (42) | 2220 (44)
  Cycle 2: number analyzed (Participants) | 63 | 68
  Cycle 2 | 11600 (36) | 35400 (49)
  Steady State (Cycle 6-10): number analyzed (Participants) | 47 | 38
  Steady State (Cycle 6-10) | 25300 (57) | 70100 (52)

11. Secondary Outcome: Number of Participants Developing Anti-tabalumab Antibodies
Time Frame: Baseline through Cycle 8
Population: Zero participants analyzed, no data collected due to compound termination.
Arm/Group | 100 mg Tabalumab+Dexamethasone+Bortezomib | 300 mg Tabalumab+Dexamethasone+Bortezomib | Placebo Comparator: Placebo + Dexamethasone + Bortezomib
Number analyzed (Participants) | 0 | 0 | 0

12. Secondary Outcome: Participants With Best Overall Response (BOR) in Each Category
Description: Stringent Complete Response-Complete Response and normal free light chain ration and no clonal cells in bone marrow Complete Response- no monoclonal protein (mp) in blood, no serum or urine mp, less than 5% plasma cells in bone marrow Very Good Partial Response-more than 90% decrease in mp and urine protein Partial Response- over 50% decrease in serum mp Stable Disease- less than 25 percent decrease of monoclonal protein Progressive Disease- 25% increase compared to lowest value of serum mp, urine mp, no measurable mp
Time Frame: Baseline to Objective Disease Progression or Initiation of New Cancer Treatment (28 Months)
Population: All randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | 100 mg Tabalumab+Dexamethasone+Bortezomib | 300 mg Tabalumab+Dexamethasone+Bortezomib | Placebo Comparator: Placebo + Dexamethasone + Bortezomib
Number analyzed (Participants) | 74 | 74 | 72
Participants
  Stringent Complete Response | 1 | 0 | 2
  Complete Response | 10 | 4 | 4
  Very Good Partial Response | 10 | 16 | 9
  Partial Response | 23 | 23 | 29
  Minimal Response | 6 | 8 | 6
  Stable Disease | 14 | 10 | 12
  Progressive Disease | 6 | 7 | 6

13. Secondary Outcome: Number of Participants With a Given Best Objective Myeloma Response (Quality of Response [QoR])
Description: Response categories in order of decreasing quality are: Stringent Complete Response(sCR),Complete Response(CR), Very Good Partial Response(VGPR),Partial Response(PR),Minimal Response(MR),Stable Disease(SD), or Progressive Disease(PD), according to the International Uniform Response Criteria for Multiple Myeloma.SCR:normal free light chain ration and no clonal cells in bone marrow;CR-no monoclonal protein(mp) in blood, no serum/urine,<5% plasma cells in bone marrow; VGPR-more than 90% decrease in mp and urine protein; PR->50% decrease in serum MP;SD-<25% decrease in mp; PD-25% increase compared to lowest value of serum mp, urine mp and no measurable mp.
Time Frame: Baseline to Objective Disease Progression or Initiation of New Cancer Treatment (up to 28 Months)
Population: All randomized participants.
Measure: Number; unit: participants
Groups:
- Placebo Comparator: Placebo + Dexamethasone + Bortezombib: Placebo administered once IV on Day 1 every 21 days for 8 cycles.Placebo administered once IV on Day 1 every 21 days for 8 cycles.
  Dexamethasone 20 mg administered once orally on Days 1, 2, 4, 5, 8, 9, 11 and 12 every 21 days for 8 cycles.
  Bortezomib 1.3 mg/m^2 administered once SQ on Days 1, 4, 8 and 11 every 21 days for 8 cycles.
Arm/Group | 100 mg Tabalumab+Dexamethasone+Bortezomib | 300 mg Tabalumab+Dexamethasone+Bortezomib | Placebo Comparator: Placebo + Dexamethasone + Bortezombib
Number analyzed (Participants) | 74 | 74 | 72
participants
  Stringent Complete Response | 1 | 0 | 2
  Complete Response | 10 | 4 | 4
  Very Good Partial Response | 10 | 16 | 9
  Partial Response | 23 | 23 | 29
  Minimal Response | 6 | 8 | 6
  Stable Disease | 14 | 10 | 12
  Progressive Disease | 6 | 7 | 6
Statistical Analysis 1: Comparison: 100 mg Tabalumab+Dexamethasone+Bortezomib vs Placebo Comparator: Placebo + Dexamethasone + Bortezombib; 100 mg Tabalumab+Dexamethasone+Bortezomib compared with Placebo Comparator: Placebo + Dexamethasone + Bortezombib, only tabalumab odds ratio compared to placebo; Test type: Superiority; p = 0.401, Regression, Logistic; Odds Ratio (OR) = 1.98
Statistical Analysis 2: Comparison: 300 mg Tabalumab+Dexamethasone+Bortezomib vs Placebo Comparator: Placebo + Dexamethasone + Bortezombib; 300 mg Tabalumab+Dexamethasone+Bortezomib compared with Placebo Comparator: Placebo + Dexamethasone + Bortezombib, only tabalumab odds ratio compared to placebo; Test type: Superiority; p = 0.455, Regression, Logistic; Odds Ratio (OR) = 1.84
Statistical Analysis 3: Comparison: 100 mg Tabalumab+Dexamethasone+Bortezomib vs 300 mg Tabalumab+Dexamethasone+Bortezomib vs Placebo Comparator: Placebo + Dexamethasone + Bortezombib; 100 mg Tabalumab+Dexamethasone+Bortezomib and 300 mg Tabalumab+Dexamethasone+Bortezomib compared with Placebo Comparator: Placebo + Dexamethasone + Bortezombib, only compared to placebo; Test type: Superiority; p = 0.419, Regression, Logistic; Odds Ratio (OR) = 1.90

14. Secondary Outcome: Overall Response Rate (ORR)
Description: Overall Response Rate (ORR) is the percentage of participants that had a response.
Time Frame: Baseline to Objective Disease Progression or Initiation of New Cancer Treatment (28 Months)
Population: All randomized participants who had a partial response or greater.
Measure: Number; unit: percentage of participants
Arm/Group | 100 mg Tabalumab+Dexamethasone+Bortezomib | 300 mg Tabalumab+Dexamethasone+Bortezomib | Placebo Comparator: Placebo + Dexamethasone + Bortezomib
Number analyzed (Participants) | 74 | 74 | 72
percentage of participants | 58.1 | 59.5 | 61.1

ADVERSE EVENTS:
Description: All randomized participants who received at least 1 dose of study drug.
Arm/Group | 100 mg Tabalumab+Dexamethasone+Bortezomib | 300 mg Tabalumab+Dexamethasone+Bortezomib | Placebo Comparator: Placebo + Dexamethasone + Bortezomib
Serious Adverse Events (participants affected / at risk) | 33/73 | 35/74 | 26/72
Other Adverse Events (participants affected / at risk) | 71/73 | 70/74 | 69/72
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 100 mg Tabalumab+Dexamethasone+Bortezomib (N=73) | 300 mg Tabalumab+Dexamethasone+Bortezomib (N=74) | Placebo Comparator: Placebo + Dexamethasone + Bortezomib (N=72)
Anaemia (Blood and lymphatic system disorders) | 2 (3) | 2 (2) | 2 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 3 (3) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 3 (3) | 1 (1) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (2) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (6) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (2) | 1 (2) | 0 (0)
Ventricular dysfunction (Cardiac disorders) | 1 (2) | 0 (0) | 0 (0)
Left ventricle outflow tract obstruction (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 2 (2) | 1 (1)
Gastric perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Ileus paralytic (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Intestinal ischaemia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Large intestinal haemorrhage (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0)
Melaena (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 1 (1)
Disease progression (General disorders) | 1 (2) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1)
General physical health deterioration (General disorders) | 2 (3) | 1 (1) | 1 (1)
Localised oedema (General disorders) | 0 (0) | 0 (0) | 1 (1)
Multi-organ failure (General disorders) | 2 (2) | 1 (1) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 1 (3)
Pyrexia (General disorders) | 1 (1) | 2 (2) | 2 (2)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Brain abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Bronchopneumonia (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Cytomegalovirus colitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Helicobacter infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 2 (2) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Infectious colitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Lobar pneumonia (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 1 (2) | 0 (0)
Otitis media (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumococcal sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumocystis jiroveci pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 9 (11) | 3 (3) | 5 (5)
Pneumonia haemophilus (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Respiratory syncytial virus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Sepsis (Infections and infestations) | 2 (3) | 5 (5) | 0 (0)
Septic shock (Infections and infestations) | 4 (8) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Soft tissue infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (3) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Multiple fractures (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Traumatic haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 1 (1) | 1 (1)
Renal function test abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1)
Troponin increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypovolaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Hepatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Plasma cell leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 1 (2)
Altered state of consciousness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Autonomic neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Loss of consciousness (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 2 (3)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0) | 2 (2)
Renal failure acute (Renal and urinary disorders) | 3 (3) | 4 (4) | 5 (5)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
Haemorrhage (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hypovolaemic shock (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
Shock haemorrhagic (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | 100 mg Tabalumab+Dexamethasone+Bortezomib (N=73) | 300 mg Tabalumab+Dexamethasone+Bortezomib (N=74) | Placebo Comparator: Placebo + Dexamethasone + Bortezomib (N=72)
Anaemia (Blood and lymphatic system disorders) | 25 (52) | 13 (25) | 17 (24)
Neutropenia (Blood and lymphatic system disorders) | 6 (8) | 4 (11) | 6 (6)
Thrombocytopenia (Blood and lymphatic system disorders) | 16 (34) | 8 (26) | 23 (60)
Atrial fibrillation (Cardiac disorders) | 4 (4) | 2 (2) | 3 (3)
Vision blurred (Eye disorders) | 2 (2) | 1 (1) | 4 (4)
Abdominal distension (Gastrointestinal disorders) | 8 (13) | 5 (5) | 5 (8)
Abdominal pain (Gastrointestinal disorders) | 5 (8) | 6 (6) | 5 (6)
Abdominal pain upper (Gastrointestinal disorders) | 5 (5) | 4 (4) | 3 (4)
Constipation (Gastrointestinal disorders) | 19 (31) | 26 (32) | 23 (30)
Diarrhoea (Gastrointestinal disorders) | 28 (44) | 27 (40) | 21 (27)
Dyspepsia (Gastrointestinal disorders) | 5 (5) | 7 (9) | 8 (10)
Nausea (Gastrointestinal disorders) | 15 (19) | 11 (12) | 14 (18)
Stomatitis (Gastrointestinal disorders) | 1 (2) | 5 (5) | 3 (3)
Toothache (Gastrointestinal disorders) | 4 (4) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 6 (7) | 5 (8) | 9 (9)
Asthenia (General disorders) | 7 (11) | 6 (6) | 9 (9)
Face oedema (General disorders) | 1 (2) | 4 (4) | 2 (2)
Fatigue (General disorders) | 28 (38) | 27 (49) | 26 (47)
Injection site erythema (General disorders) | 4 (4) | 2 (5) | 1 (1)
Injection site reaction (General disorders) | 6 (13) | 3 (5) | 3 (7)
Oedema (General disorders) | 1 (5) | 4 (35) | 4 (25)
Oedema peripheral (General disorders) | 14 (57) | 15 (69) | 8 (27)
Pain (General disorders) | 6 (7) | 3 (3) | 2 (3)
Pyrexia (General disorders) | 11 (13) | 10 (13) | 6 (8)
Herpes zoster (Infections and infestations) | 4 (4) | 6 (7) | 4 (5)
Nasopharyngitis (Infections and infestations) | 3 (5) | 4 (4) | 2 (2)
Pneumonia (Infections and infestations) | 6 (7) | 3 (4) | 3 (3)
Respiratory tract infection (Infections and infestations) | 8 (14) | 3 (4) | 0 (0)
Sinusitis (Infections and infestations) | 3 (3) | 4 (4) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 11 (17) | 18 (31) | 20 (27)
Urinary tract infection (Infections and infestations) | 8 (12) | 4 (4) | 5 (5)
Contusion (Injury, poisoning and procedural complications) | 3 (3) | 5 (5) | 2 (3)
Alanine aminotransferase increased (Investigations) | 8 (11) | 6 (6) | 1 (2)
Aspartate aminotransferase increased (Investigations) | 7 (9) | 6 (6) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 3 (5) | 4 (5) | 0 (0)
Blood cholesterol increased (Investigations) | 5 (12) | 2 (6) | 6 (10)
Lymphocyte count decreased (Investigations) | 1 (1) | 5 (13) | 1 (1)
Neutrophil count decreased (Investigations) | 4 (8) | 2 (3) | 1 (5)
Platelet count decreased (Investigations) | 16 (46) | 7 (10) | 8 (15)
Weight decreased (Investigations) | 5 (7) | 8 (11) | 5 (5)
Weight increased (Investigations) | 4 (4) | 3 (3) | 3 (5)
Decreased appetite (Metabolism and nutrition disorders) | 12 (13) | 12 (13) | 8 (10)
Dehydration (Metabolism and nutrition disorders) | 3 (5) | 1 (1) | 5 (7)
Hyperglycaemia (Metabolism and nutrition disorders) | 5 (11) | 5 (10) | 7 (11)
Hyperkalaemia (Metabolism and nutrition disorders) | 3 (3) | 1 (1) | 5 (7)
Hypocalcaemia (Metabolism and nutrition disorders) | 7 (12) | 7 (9) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 7 (12) | 7 (8) | 3 (3)
Hyponatraemia (Metabolism and nutrition disorders) | 3 (3) | 4 (4) | 3 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (5) | 7 (7) | 3 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 7 (10) | 12 (14) | 13 (16)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 6 (7) | 4 (5) | 6 (9)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 7 (8) | 0 (0) | 4 (4)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 4 (5) | 4 (5)
Myalgia (Musculoskeletal and connective tissue disorders) | 6 (7) | 3 (3) | 5 (7)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 (11) | 10 (14) | 11 (11)
Dizziness (Nervous system disorders) | 6 (7) | 15 (20) | 16 (23)
Dysgeusia (Nervous system disorders) | 5 (5) | 3 (4) | 2 (2)
Headache (Nervous system disorders) | 9 (10) | 3 (4) | 5 (9)
Hypoaesthesia (Nervous system disorders) | 4 (5) | 0 (0) | 1 (1)
Neuralgia (Nervous system disorders) | 1 (1) | 9 (12) | 7 (10)
Neuropathy peripheral (Nervous system disorders) | 17 (20) | 11 (16) | 13 (25)
Paraesthesia (Nervous system disorders) | 8 (12) | 8 (11) | 5 (6)
Peripheral sensory neuropathy (Nervous system disorders) | 10 (16) | 19 (32) | 17 (31)
Tremor (Nervous system disorders) | 4 (4) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 5 (5) | 4 (4)
Insomnia (Psychiatric disorders) | 12 (12) | 15 (19) | 11 (24)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 2/29 (2) | 0/37 (0) | 1/40 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 8 (9) | 16 (17) | 13 (18)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9 (10) | 8 (8) | 11 (16)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 (8) | 3 (3) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 5 (8) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 5 (6) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 7 (16) | 7 (16) | 2 (6)
Orthostatic hypotension (Vascular disorders) | 3 (4) | 4 (5) | 5 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days